CLINICAL TRIAL: NCT05917587
Title: Metformin for the Treatment of Microvascular Dysfunction After Gestational Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202303345; 1R01HL169201-01 (NIH)
Record Dates: First submitted 2023-06-06; First posted 2023-06-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; postpartum; vascular
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Active Comparator)
  Interventions: Drug: Metformin Hydrochloride
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — 12 weeks: 850mg metformin once daily for first 7 days then twice daily for the remaining 11 weeks.
  Arms: metformin
Other: placebo — 12 weeks: placebo tablet once daily for the first 7 days then twice daily for the remaining 11 weeks.
  Arms: placebo

SUMMARY:
The purpose of this investigation is to examine the mechanisms mediating vascular dysfunction in women who have had gestational diabetes and how metformin may be a valuable treatment tool to improve microvascular function in these women before the onset of disease.

DETAILED DESCRIPTION:
Women with a history of gestational diabetes mellitus (GDM) are at a 2-fold greater risk for the development of overt cardiovascular disease (CVD) following the effected pregnancy. While subsequent development of type II diabetes elevates this risk, prior GDM is an independent risk factor for CVD morbidity, particularly within the first decade postpartum. GDM is associated with impaired endothelial function during pregnancy and decrements in macro- and microvascular function persist postpartum, despite the remission of insulin resistance following delivery. Collectively, while the association between GDM and elevated lifetime CVD risk is clear, and available evidence demonstrates a link between GDM and vascular dysfunction in the decade following pregnancy, the mechanisms mediating this persistent dysfunction remain unexamined.

The purpose of this investigation is to examine the mechanisms mediating vascular dysfunction in women who have had gestational diabetes and how metformin may be a valuable treatment tool to improve microvascular function in these women before the onset of disease. This study will give rise to a new line of research that will center around the goal of improving lifetime cardiovascular outcomes in women with a history of GDM.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) they examine the blood vessels in a dime-sized area of the skin in women who have had GDM. Local heating of the skin at the microdialysis sites is used to explore differences in mechanisms governing microvascular control. As a compliment to these measurements, the investigators also draw blood from the subjects and isolate the inflammatory cells.

ELIGIBILITY:
Inclusion Criteria:

* ≥12 weeks and ≤5 years postpartum
* history of GDM or healthy pregnancy

Exclusion Criteria:

* prediabetes or diabetes (HbA1c ≥5.7%)
* current tobacco use
* cardiovascular or metabolic disease
* cardiovascular or metabolic medication
* history of hypertension during pregnancy
* current pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
blood flow response to acetylcholine | baseline
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to acetylcholine
blood flow response to acetylcholine | 1 week of treatment
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to acetylcholine
blood flow response to acetylcholine | 6 weeks of treatment
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to acetylcholine
blood flow response to acetylcholine | 12 weeks of treatment
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to acetylcholine
blood flow response to insulin | baseline
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to insulin
blood flow response to insulin | 1 week of treatment
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to insulin
blood flow response to insulin | 6 weeks of treatment
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to insulin
blood flow response to insulin | 12 weeks of treatment
  cutaneous microvascular dilation (cutaneous conductance ; %max) response to insulin

SECONDARY OUTCOMES:
Percentage of nitric oxide-dependent dilation | baseline
  NO-dependent (%) cutaneous microvascular dilation response to acetylcholine
Percentage nitric oxide-dependent dilation | 1 week of treatment
  NO-dependent (%) cutaneous microvascular dilation response to acetylcholine
Percentage of nitric oxide-dependent dilation | 6 weeks of treatment
  NO-dependent (%) cutaneous microvascular dilation response to acetylcholine
Percentage of nitric oxide-dependent dilation | 12 weeks of treatment
  NO-dependent (%) cutaneous microvascular dilation response to acetylcholine

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Findings from the primary studies will be published and submitted to PubMed Central in compliance with the NIH public access policy. These findings will also be made public through the clinicaltrial.gov record. The final data set will be stripped of any identifying data prior to release for sharing. We will make the data and any associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using the data only for research purposes and not to identify any one individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after all analyses are completed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code